CLINICAL TRIAL: NCT01244503
Title: Prediction of Severity of Liver Disease in Patients With Suspected Nonalcoholic Fatty Liver Disease (NAFLD) by 13C Octanoate Breath Test (OBT)
Brief Title: Prediction of Severity of Liver Disease by a 13C Octanoate Breath Test (OBT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Budgetary Issues
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NASH-BID-FIS-808
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Metabolic Syndrome; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease | interventions — octanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium Octanoate Breath Test (Experimental): Only subjects with metabolic syndrome and suspected non alcoholic fatty liver disease will undergo breath test. They must not have any other liver disease.
  Interventions: Drug: Sodium Octanoate Breath Test

INTERVENTIONS:
Drug: Sodium Octanoate Breath Test — 100 mg of 13-C labeled sodium octanoate (Octanoate for short) is to be dissolved in 1 cup of tap water and administered to subject after baseline breath collection is completed.
  Other Names: Octanaote, sodium octanoate

SUMMARY:
The purpose of the study is to demonstrate that the ¹³C-Octanoate Breath Test (OBT) can be used as an aid, in conjunction with other clinical information and medical history, for evaluating disease severity and detecting NASH with a high probability.

DETAILED DESCRIPTION:
The OBT was chosen to assess, along with other parameters, liver health in subjects suspected of NAFLD (non alcoholic fatty liver disease).

Octanoate is absorbed promptly from the intestinal lumen and transported rapidly to the liver through the portal venous system, enters the hepatic mitochondria independently of the carnitine transport system and undergoes hepatic mitochondrial beta-oxidation which produces acetyl coenzyme A (CoA). Finally, acetyl CoA enters the Krebs cycle and is oxidized by carbon dioxide (CO2). This is a non invasive test that can be performed routinely at every visit to assess disease severity. The subject is connected to a breath analyzer via a nasal cannula for approximately 1 hour, that measures baseline breath and changes in delta over baseline due to metabolization of Octanoate.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women (>18 years of age)
* • Liver -biopsy ( at least 1.7 cm and 4 portal tracts) performed within 6 months of breath test or planned within the next 6 weeks, providing no treatment for liver disease was given between the biopsy and the OBT Any elevation of liver enzymes above the upper limit of normal (any or all of the following: AST,ALT, GGT, Alkaline phosphatase)
* At least one of the features of the metabolic syndrome

  * waist circumference > 100 cm for men, 88 cm for women
  * triglycerides > 150 mg/dl
  * fasting blood sugar > 110 mg/dl
  * HDL cholesterol < 40 mg/dl
  * blood pressure > 130/85 mm Hg
* No other known co-existent liver disease, excluded by appropriate serologic testing

Exclusion Criteria:

* Positive studies for any of the following:
* hepatitis C (PCR)
* hepatitis B (surface antigen or DNA)
* iron saturation > 60% + gene test for hereditary hemochromatosis
* antinuclear antibody at a titer > 1: 160 along with hypergammaglobulinemia and ALT levels>250 U/L

  * Patient has Alpha-1-antitrypsin level below lower limit of normal (< 150 mg/dl)
  * Patient has alcohol consumption > 20 gm/day for women and > 30 gm/day for men
  * Patient is pregnant
  * Patient has been taking known hepatotoxic drugs e.g. (e.g.acebutolol, indomethacin,phenylbutazone,allopurinol,isoniazid,phenytoin,atenolol,ketoconazole,piroxicam,carbamazepine,labetalol,probenecid,cimetidine,maprotiline,pyrazinamide,dantrolene, metoprolol,quinidine,diclofenac, mianserin)• Patients that have had more than 10% reduction in body weight since biopsy
  * Patient with known severe congestive heart failure (LVEF on echocardiogram < 20%)
  * Patient with known severe pulmonary hypertension (By echocardiogram, PAS >45 mmHg)
  * Patient with uncontrolled diabetes mellitus (HA1c>10)
  * Patient with previous surgical bypass surgery
  * Patient with extensive short bowel syndrome(>100 cm)
  * Patient currently receiving total parenteral nutrition
  * Patient is a recipients of any organ transplant
  * Patients that received any anti-viral treatment or any other liver therapy between the time of the biopsy and the breath test.
  * Women who are pregnant
  * Patients with an acute current exacerbation of chronic obstructive pulmonary disease or bronchial asthma.
  * Patient has taken drugs that can interfere with octanoate metabolism or can also cause NAFLD independent of the metabolic syndrome, including: corticosteroids, amiodarone, tetracycline, valproic acid, methotrexate, stavudine, zidovudine.
  * Patients unable or refuse to sign informed consent
  * Patients that based on the opinion of the investigator should not be enrolled into this study
  * Patients that are participating in other clinical trials evaluating experimental treatments or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun J. Sanyal, M.D., Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Octanoate Breath Test
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only subjects with metabolic syndrome and suspected non alcoholic fatty liver disease will undergo breath test. They must not have any other liver disease.
Arm/Group | Sodium Octanoate Breath Test
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 57
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 54
  Israel | 7
Blood pressure diastolic [Mean (Standard Deviation); unit: mmHg] | 75 (10)
Blood pressure systolic [Mean (Standard Deviation); unit: mmHg] | 135 (18)
Weight [Mean (Standard Deviation); unit: Kg] | 100 (22)
Height [Mean (Standard Deviation); unit: centimeters] | 167 (21)

OUTCOME MEASURES:

1. Primary Outcome: The Peak Value of the PDR (Percentage Dose Recovery of 13C) of OBT (Octanoate Breath Test)
Description: To assess the ability of the OBT to assess disease severity in patients with suspected NAFLD (non alcoholic fatty liver disease) compared to NAS (Non-alcoholic-steatohepatitis (NASH) Activity Score) scoring system, where steatosis is scaled from 0-3, lobular inflammation is scaled from 0-3 and hepatocellular ballooning is scaled from 0-2. NAS score greater or equal to 5 indicates NASH. The higher the PDR peak, the better the liver health and function.PDR units are percent per hour of 13C dose recovery and describes rate of metabolism. The PDR peak is the highest rate of metabolism the liver reaches.The total range of NAS is 0-8.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: PDR peak value (%/hour)
Arm/Group | Sodium Octanoate Breath Test
Number analyzed (Participants) | 61
PDR peak value (%/hour) | 23.27 (4.93)

2. Secondary Outcome: Histology -NAS Scoring of Liver Biopsy
Description: OBT will be compared to histology (including NAS score as described above)and other parameters to develop severity score. Only subjects with biopsy from routine clinical practice will be enrolled.
  NAS (Non-alcoholic-steatohepatitis (NASH) Activity Score) scoring system includes the following components: steatosis, which is scaled from 0-3, lobular inflammation, which is scaled from 0-3 and hepatocellular ballooning, which is scaled from 0-2. NAS score greater or equal to 5 indicates NASH. The range of the NAS score is from 0-8.
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sodium Octanoate Breath Test
Number analyzed (Participants) | 61
units on a scale | 3.71 (1.60)

ADVERSE EVENTS:
Description: No breath test related adverse events were reported
Arm/Group | Sodium Octanoate Breath Test
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 4/61
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Octanoate Breath Test (N=61)
Pain (General disorders) | 1 (1) — Upper right quadrant pain
Lightheadedness (General disorders) | 1 (1) — Non liver related
Hyperglycemia (Endocrine disorders) | 1 (1)
Odiferous breath (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days